CLINICAL TRIAL: NCT03311789
Title: A Pilot Study of PD-1 Inhibitor in Combination With Gemcitabine/Cisplatin for Patients With Advanced Unresectable or Metastatic Biliary Tract Cancers
Brief Title: Study of PD-1 Inhibitor in Combination With Gemcitabine/Cisplatin for Advancer BTCs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Ph.D, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-024
Record Dates: First submitted 2017-10-04; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Immune Checkpoint Inhibitors; Gemcitabine; Cisplatin; Nivolumab; camrelizumab

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be treated with PD-1 inhibitor in combination with gemcitabine/cisplatin chemotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 inhibitor + Gemcitabine+Cisplatin (Experimental): Patients will be enrolled in the experimental arm and will receive Gemcitabine on day 1 and 5 (1000mg/m2 ) +Cisplatin on day 1(75mg/m2)+ PD-1 inhibitor on day 3 (Nivolumab 3mg/kg, or SHR-1210 200mg) every 3 weeks. If there is continued benefit after 6 months, PD-1 inhibitor will be administered as maintenance treatment until tumor progression or death.
  Interventions: Drug: PD-1 inhibitor + Gemcitabine + Cisplatin

INTERVENTIONS:
Drug: PD-1 inhibitor + Gemcitabine + Cisplatin — Gemcitabine: 1000mg/m2 on day 1 and 5 every 3 weeks. Cisplatin: 75mg/m2 on day 1 every 3 weeks. PD-1 inhibitor: Nivolumab 3mg/kg, or SHR-1210 200mg.
  Other Names: Nivolumab or SHR-1210

SUMMARY:
This is a single-arm, phase I/II trial in biliary tract cancer (BTC) patients. The purpose of this trial is to evaluate the safety and effect of PD-1 inhibitor in combination with gemcitabine/cisplatin chemotherapy in patients with advanced unresectable or metastatic BTCs.

The primary objective: 6-month progression free survival (PFS). The second objectives: objective clinical response(according to RECIST version 1.1), safety, symptom control and quality of life (QoL) (according to EORTC QoL C30 and BIL 21), overall survival. The exploratory objectives: assessment of immunological response (cytokines, lymphocyte phenotype, immunoglobulins), and evaluation of pathological, immunological and clinical predictive factors for response/toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years with estimated life expectancy >3 months.
* Histopathological/cytological diagnosis of unresectable or recurrent / metastatic biliary tract carcinoma (intra-hepatic, extrahepatic or gall bladder) and had at least one measurable disease (≥1cm) by CT or MRI.
* Patients should provide samples of tumor tissue biopsied or resected no more than 3 months before enrollment and be willing to accept biopsy in the process of the study.
* Patients may have received prior radiotherapy,chemotherapy,or other local ablative therapies, which completed ≥ 4 weeks prior to registration AND patient has recovered to <= grade 1 toxicity.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-2.
* Adequate organ and marrow function obtained ≤ 2 weeks prior to registration as defined below:

leukocytes greater than or equal to 3.0 x 10^9/L absolute neutrophil count greater than or equal to 1.0 x 10^9/L platelets greater than or equal to 100 x 10^9/L hemoglobin greater than or equal to 90 g/L total bilirubin less than or equal to 2 xULN serum albumin should be no less than 25g/L ALT or AST less than 2 xULN serum creatinine less than 1.5 x ULN

* Ability to understand and willingness to sign a written informed consent document.
* women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and up to 120 days after the last dose of the drug.

Exclusion Criteria:

* Active, known or suspected autoimmune diseases.
* Known brain metastases or active central nervous system (CNS). If patients with CNS metastases were treated with radiotherapy for at least 3 months prior to enrollment and have no central nervous symptoms and are off corticosteroids, they will be eligible but will need a Brain MRI prior to enrollment.
* Participants are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
* Prior therapy with anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody (including ipilimumab or any other antibody specifically targeting T-cell costimulation or checkpoint pathways).
* History of severe hypersensitive reactions to other monoclonal antibodies.
* History of allergy or intolerance to study drug components.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
* Uncontrolled intercurrent illness including ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
* History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
* Pregnant or breast-feeding patients. Women of childbearing potential must have a pregnancy test performed within 7 days before the enrollment, and a negative result must be documented.
* Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Vaccination within 30 days of study enrollment.
* Active bleeding or known hemorrhagic tendency.
* Patients with unhealed surgical wounds for more than 30 days.
* Being participating any other trials or withdraw within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients alive and without progression at 6 months | 6 months
  The primary objective of this trial is the progression free survival (PFS) at 6 months in patients with advanced unresectable or metastatic BTCs treated with PD-1 inhibitor in combination with gemcitabine plus cisplatin. Progression will be defined clinically or on imaging as per immune related response evaluation criteria in solid tumors (irRECIST) definition

SECONDARY OUTCOMES:
The percentage of patients that respond to combination treatment | Enrolled patients will be followed until death, withdrawal from study, or until 2 years.
  Overall response rate is defined as the sum of partial responses and complete responses. Partial and complete response will be defined as per irRECIST criteria.
Median overall survival time | Patients will be followed until death, withdrawal from study, or until 2 years.
  The median overall survival (OS) time is defined as the time from enrollment to death.
List of adverse event frequency and grade | Up to 120 days after last administration of PD-1 inhibitor
  To evaluate the safety of PD-1 inhibitor in combination with standard chemotherapy in patients with advanced BTCs according to CTCAE 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Study Director — Department of Biotherapeutic, Chinese PLA General Hospital
Locations (1):
- Department of Biotherapeutic, Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng K, Liu Y, Zhao Y, Yang Q, Dong L, Liu J, Li X, Zhao Z, Mei Q, Han W. Efficacy and biomarker analysis of nivolumab plus gemcitabine and cisplatin in patients with unresectable or metastatic biliary tract cancers: results from a phase II study. J Immunother Cancer. 2020 Jun;8(1):e000367. doi: 10.1136/jitc-2019-000367. PMID 32487569